CLINICAL TRIAL: NCT03001232
Title: Enriched Environment and Dementia: The Effect of an Individual Daily Calendar on the Activity Level and Mental Functions of Persons With Dementia in a Nursing Home
Brief Title: The Effect of Movement-oriented Dementia Care on ADL and QoL of Dementia Patients in Nursing Homes
Acronym: Solis MDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Zorggroep Solis (Unknown)
Responsible Party: Principal Investigator, Marinda Henskens, Msc, VU University of Amsterdam
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: METc Vumc: 2013.311/A2015.245
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-01

CONDITIONS: Dementia
Keywords: Movement-oriented Dementia Care; QoL; ADL; Nursing Home
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Movement-oriented Dementia Care (Experimental): The experimental group received movement-oriented dementia care for a period of twelve months.Movement-oriented dementia care is a multidisciplinary approach in which all involved disciplines focus on stimulating physical activity and independence as much as possible. This way physical activity is stimulated at all times for the participants.
  Interventions: Behavioral: Movement-oriented Dementia Care
- Care as usual (No Intervention): The control group received care as usual

INTERVENTIONS:
Behavioral: Movement-oriented Dementia Care — The intervention is a new multidisciplinary approach that focuses on optimizing physical activity and independence in daily care and activities. MDC intended to incorporate all persons surrounding the patients. The nursing staff was intensively trained by an expert in MDC, and played a central role in continuously stimulating patients to function as independently as possible. Geriatric physicians and physiotherapists advised the nursing staff about participants' medical and physical limitations to ensure safe stimulation. Consequently, a plan was created for each resident to determine the daily routines they were capable of performing themselves. Caregivers and volunteers were informed about the benefits of an active lifestyle during several open meetings.
  Arms: Movement-oriented Dementia Care

SUMMARY:
The purpose of this study is to determine whether movement-oriented dementia care has a positive effect on quality of life and independence in activities of daily living (ADL) in nursing-home residents with dementia.

It was hypothesized that movement-oriented dementia care has a positive effect on quality of life and independence in ADL, as well as on mood, behavior, cognition and physical functioning, in comparison to regular care.

DETAILED DESCRIPTION:
Background:

In the Netherlands, an estimated number of 70.000 patients with dementia are institutionalized. This number is expected to increase rapidly in the coming years due to the aging population. Loss of independence in activities of daily living (ADL) is an important predictor for institutionalization and an important determinant for the quality of life. Once institutionalized, independence in ADL tends to decline even more rapid.This rapid decline may be due to insufficient stimulation of the patients' remaining abilities. Underestimating the patient's abilities may contribute to the inactive lifestyle in nursing homes. An inactive lifestyle negatively affects multiple disease outcomes. In the present study, movement-oriented dementia care (MDC) is implemented on psychogeriatric wards of a Dutch nursing home. MDC focuses on the integration of physical activity in the daily lives of nursing home residents with dementia. The key element of MDC is the multidisciplinary approach to ensure physical stimulation at all times. The following disciplines are involved in MDC: nursing staff, department heads, paramedics (physiotherapists and occupational therapists), psychologists, geriatrics specialists, activity leaders, volunteers and family caregivers. The primary aim is to evaluate the effect of MDC on ADL independence and quality of life. Additionally, the effect on mood, behaviour, cognition, and physical fitness is investigated.

The present study was a non-randomized 12-month longitudinal study with two parallel groups. The study was approved by the Medical Ethical Exam Committee (METc) of the VUmc.

Participants were residents from five psychogeriatric wards of two locations of nursing home Solis in Deventer. All participants were diagnosed with dementia.

Recruitment: In the first place, the staff of Nursing home Solis was informed about the intervention. Consequently, an initial selection of suitable clients took place. Clients receiving palliative care did not participate in the study. Suitable clients and their caregivers were informed about the study by means of an informative presentation as well as an informative letter in which clients and their caregivers were asked to give informed consent.

Randomisation:Two locations of nursing home Solis were non-randomly allocated to the experimental or control condition. Participants living at the experimental location received movement-oriented dementia care (MDC), while participants living at the control location received care as usual.

Procedure: Movement-oriented Dementia Care was given to as many residents as possible from the psychogeriatric wards of the intervention location. In order to properly implement movement-oriented care, nursing staff, activity leaders and living room staff were offered a schooling aimed at increasing awareness of the importance of movement, as well as providing tools for stimulating movement in elderly with dementia. Caregivers and volunteers received information about movement during an information meeting. The execution of the movement-oriented care differed per discipline. Nursing staff continuously encouraged clients to function as independently as possible. This regards activities such as getting dressed, preparing meals, pouring coffee, and toilet use. Paramedics coached the nursing staff by specifying medical and physical limits of each participant. Additionally, they gave advice on how to handle specific situations. They also informed and coached caregivers on how to safely stimulate movement with clients. Based on these advises, a plan was created for each resident to determine the daily routines that they are capable of performing, as well as how to stimulate the participants to engage in physical activities. Activity leaders were informed on how to include movement interventions in their activities. In addition, activity leaders constructed a leisure-care calendar focusing on general activities based on personal preferences and potentials. Family caregivers and volunteers were encouraged to stimulate physical activity of the patients in general.

Nursing staff were trained by an expert in MDC (three sessions of three hours), in order to increase awareness of the importance of physical activity, as well as the role of physical activity in ADL. Additionally, paramedics received a two-hour meeting informing them on their role in advising nursing staff. Volunteers and family caregivers were informed about the benefits of an active lifestyle during several open meetings.

The outcome variables were measured 5 times, i.e. at baseline and after 3, 6, 9, and 12 months of the intervention. Trained physiotherapists performed the measurements with participants, while nursing staff and caregivers were asked to fill in questionnaires. The test battery administered by the clients had a maximum duration of 30 to 45 minutes, in which the client was free to take breaks.

To ensure compliance to the intervention, one staff member at each psychogeriatric ward became an 'ambassador' of MDC, responsible for implementation at their ward. Process evaluations were administered for nursing staff and caregivers every three months to measure the extent of implementation. These process evaluations consisted of structured interviews and questionnaires. Questionnaires were completed by nursing staff and family caregivers every three months. Structured interviews were conducted with members of a multidisciplinary focus group after three and nine months. The focus group consisted of 12 professionals; nurses, activity leaders, heads of the departments, 'ambassadors', a physiotherapist and an occupational therapist. The process evaluations focused on the following elements:

* To which extent did staff and family carers prepare to provide MDC?
* Which aspects of MDC are applied?
* Is MDC applied according to its core principles?
* To what extent are participants stimulated to be physically active?
* Are the staff and family carers satisfied with the execution of MDC?
* What barriers are experienced?

The following demographic data was registered per participant: subtype dementia, birth year (age), sex, education, severity of dementia, comorbidities, cardiovascular risk factors and medication use.

The severity of dementia was determined using the Mini Mental State Examination (MMSE). The scores ranged from 0 (severe cognitive impairment) to 30 (no cognitive impairment). The recommended cut-off point of 24 was applied, with a score of 23 or lower indicating dementia.

Comorbidities were derived from the medical charts of the participants and were categorized according to the Dutch translation of the Long-Term Care Facility Resident Assessment Instrument (RAI), section I disease diagnosis. The section consists of 44 subcategories that belong to eight categories. The sum of the subcategories was used as a comorbidity score. Information regarding cardiovascular risk factors was derived from the medical charts of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia (based on medical charts)
* Living in a psychogeriatric ward of Solis for at least three weeks
* 65 years of age or older

Exclusion Criteria:

* Very bad vision
* Psychotic symptoms
* A palliative care protocol
* A score on the Mini-Mental State Examination (MMSE) of 25 or higher

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Activities of Daily Living (ADL), measured with the Barthel Index. | baseline and 3, 6, 9 and 12 months after baseline assessment
  The Barthel Index is a survey consisting of 10 performance items (e.g. toilet use, dressing) rated on an ordinal scale (two-point, three-point or four-point scale), indicating the level of help needed. Scores range from 0 to 20, with higher scores representing a higher level of functional independence.
Change from Baseline in Quality of Life (QoL), measured with the Qualidem | baseline and 3, 6, 9 and 12 months after baseline assessment
  The Qualidem is a questionnaire with 40 items of observable behaviour rated on a four-point rating scale, ranging from 1 (never) to 4 (often). There is no total score; scores can only be obtained for the nine subscales. For each subscale, a higher score represented a better quality of life.

SECONDARY OUTCOMES:
Change from Baseline in general cognitive functions, measured with the Severe Impairment Battery 8 (SIB-8). | baseline and 3, 6, 9 and 12 months after baseline assessment.
  The SIB-8 consists of eight questions measuring orientation in time, writing, fluency, naming, and attention. Scores range from 0 to 16, with higher scores indicating better cognitive functions
Change from Baseline in mood, measured with the Cornell Scale for Depression in Dementia (CSDD). | baseline and 3, 6, 9 and 12 months after baseline assessment
  The CSDD consists of 30 questions rated on a two-point scale ranging from 0 (absent) to 2 (severe). Scores range from 0 to 38, with higher scores representing a higher level of depressive symptoms.
Change from Baseline in behaviour, measured with the Apathy Evaluation Scale-10 (AES-10). | baseline and 3, 6, 9 and 12 months after baseline assessment.
  The AES-10 is a selection of 10 items from the original AES, which were applicable to nursing home residents. The items represent behaviours (contra) indicative for apathy (e.g. being motivated). Each item is rated on a four-point scale, ranging from 1 (not characteristic) to 4 (very characteristic). Scores range from 10 to 40, which higher scores representing more apathetic behaviour.
Change from Baseline in behaviour, measured with the Cohen-Mansfield Agitation Inventory (CMAI). | baseline and 3, 6, 9 and 12 months after baseline assessment.
  The CMAI is a questionnaire consisting of 29 items representing types of agitated behaviour, rated on a seven-point scale. Higher scores indicate more agitated behaviour.
Change from Baseline in aerobic fitness, measured with the two minute walking test (2mWT). | baseline and 3, 6, 9 and 12 months after baseline assessment
  The participant was requested to walk the largest distance possible during a time period of two minutes. The participant was allowed to use a walking device and take breaks if necessary.
Change from Baseline in functional mobility and fall risk, measured with the Timed up and go (TUG). | baseline and 3, 6, 9 and 12 months after baseline assessment
  The participant was asked to stand up from a chair with armrests, walk three metres, turn around, walk back to the chair, and sit down again. The participant was allowed to use a walking device. The time it took for the participant to perform these steps was recorded by the examiner.
Change from Baseline in walking speed, measured with the ten meter timed walk. | baseline and 3, 6, 9 and 12 months after baseline assessment.
  The participant was asked to walk 10 meters in a comfortable speed. The participant was allowed to use a walking device. The test was repeated three times, where the fastest attempt was used as an outcome measure for walking speed as recorded in metres per second.

OTHER OUTCOMES:
Degree of implementation of MDC at each ward measured with process evaluations. | 3, 6, 9 and 12 months of intervention.
  Process evaluations included both questionnaires and structured interviews. Questionnaires were completed by the nursing staff and family caregivers. Structured interviews were conducted with members of a multidisciplinary focus group

CONTACTS AND LOCATIONS:
Overall Officials: Marinda Henskens, Msc, Principal Investigator — VU University of Amsterdam; Erik JA Scherder, Prof. Dr., Principal Investigator — VU University of Amsterdam; Susan Vrijkotte, Msc, Study Director — Zorggroep Solis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballard C, O'Brien J, James I, Mynt P, Lana M, Potkins D, Reichelt K, Lee L, Swann A, Fossey J. Quality of life for people with dementia living in residential and nursing home care: the impact of performance on activities of daily living, behavioral and psychological symptoms, language skills, and psychotropic drugs. Int Psychogeriatr. 2001 Mar;13(1):93-106. doi: 10.1017/s1041610201007499. PMID 11352339
- [Background] Blankevoort CG, van Heuvelen MJ, Boersma F, Luning H, de Jong J, Scherder EJ. Review of effects of physical activity on strength, balance, mobility and ADL performance in elderly subjects with dementia. Dement Geriatr Cogn Disord. 2010;30(5):392-402. doi: 10.1159/000321357. Epub 2010 Oct 28. PMID 20980758
- [Background] Edwards N, Gardiner M, Ritchie DM, Baldwin K, Sands L. Effect of exercise on negative affect in residents in special care units with moderate to severe dementia. Alzheimer Dis Assoc Disord. 2008 Oct-Dec;22(4):362-8. doi: 10.1097/WAD.0b013e31818ecbbc. PMID 18978600
- [Background] Burge E, Kuhne N, Berchtold A, Maupetit C, von Gunten A. Impact of physical activity on activity of daily living in moderate to severe dementia: a critical review. Eur Rev Aging Phys Act. 2012 Apr;9(1):27-39. doi: 10.1007/s11556-011-0092-y. Epub 2011 Dec 15. PMID 22639696
- [Background] Dechamps A, Diolez P, Thiaudiere E, Tulon A, Onifade C, Vuong T, Helmer C, Bourdel-Marchasson I. Effects of exercise programs to prevent decline in health-related quality of life in highly deconditioned institutionalized elderly persons: a randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):162-9. doi: 10.1001/archinternmed.2009.489. PMID 20101011
- [Background] Kemoun G, Thibaud M, Roumagne N, Carette P, Albinet C, Toussaint L, Paccalin M, Dugue B. Effects of a physical training programme on cognitive function and walking efficiency in elderly persons with dementia. Dement Geriatr Cogn Disord. 2010;29(2):109-14. doi: 10.1159/000272435. Epub 2010 Feb 11. PMID 20150731
- [Background] Morris JN, Fiatarone M, Kiely DK, Belleville-Taylor P, Murphy K, Littlehale S, Ooi WL, O'Neill E, Doyle N. Nursing rehabilitation and exercise strategies in the nursing home. J Gerontol A Biol Sci Med Sci. 1999 Oct;54(10):M494-500. doi: 10.1093/gerona/54.10.m494. PMID 10568531
- [Background] Wetzels RB, Zuidema SU, de Jonghe JF, Verhey FR, Koopmans RT. Determinants of quality of life in nursing home residents with dementia. Dement Geriatr Cogn Disord. 2010;29(3):189-97. doi: 10.1159/000280437. Epub 2010 Mar 6. PMID 20215750
- [Background] Galik E, Resnick B, Hammersla M, Brightwater J. Optimizing function and physical activity among nursing home residents with dementia: testing the impact of function-focused care. Gerontologist. 2014 Dec;54(6):930-43. doi: 10.1093/geront/gnt108. Epub 2013 Oct 3. PMID 24092822
- [Derived] Henskens M, Nauta IM, Scherder EJA, Oosterveld FGJ, Vrijkotte S. Implementation and effects of Movement-oriented Restorative Care in a nursing home - a quasi-experimental study. BMC Geriatr. 2017 Oct 23;17(1):243. doi: 10.1186/s12877-017-0642-x. PMID 29058632